CLINICAL TRIAL: NCT05090553
Title: Cutibacterium Acnes Colonization on Intervertebral Discs of Patients With Low Back Pain: Protocol for an Analytical Study With Microbiological, Phenotypic, Genotypic and Multiomics Techniques
Brief Title: Protocol for an Analytical Study With Microbiological, Phenotypic, Genotypic and Multiomics Techniques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gaffree & Guinle Universitary Hospital (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Vinicius Magno da Rocha, Clinical Professor, Gaffree & Guinle Universitary Hospital
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: VMRDocProtocol_2021
Record Dates: First submitted 2021-09-28; First posted 2021-10-22 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Back Pain, Low; Degenerative Disc Disease
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither the patient nor the surgeons will have access to the results of microbiological cultures or molecular analysis. The radiologist who will review the exams will also be blinded to patient data and laboratory results. The researcher who will analyze the pain and function scores will also be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- surgical treatment (Active Comparator): Lumbar Spinal Fusion Surgery
  Interventions: Procedure: Lumbar Spinal Fusion Surgery
- Bacterial culture (Experimental): Cutibacterium acnes culture in two different atmosphere:
  * Carbon dioxide (CO2) from 5% up to 10%
  * CO2 10%, H2 10% and N2 80%
  Interventions: Biological: Bacterial culture
- Phenotypic and genotypic characterization (Experimental): Mass spectrometry and (Polimerase Chain Reaction) PCR
  Interventions: Genetic: Phenotypic and genotypic characterization
- Multiomics analysis (Experimental): * Genome sequencing
  * Proteomics
  * Metabolomics
  Interventions: Genetic: Multiomics analysis

INTERVENTIONS:
Procedure: Lumbar Spinal Fusion Surgery — During surgery will be collected five disc fragments and five fragments of muscle-ligament tissue adjacent to the collected disc.
  Arms: surgical treatment
Biological: Bacterial culture — Samples will be seeded on blood agar and anaerobic blood agar plates. After sowing in solid media, the swab will be inoculated in thioglycolate medium, where it will remain for 14 days
  Arms: Bacterial culture
Genetic: Phenotypic and genotypic characterization — The phenotypic identification of the species will be carried out through mass spectrometry, with the MALDI-TOF equipment.
  PCR analyzes performed in two phases, the first to confirm the presence of bacteria (target and non-target) using primers capable of amplifying eubacteria ribosomal deoxyribonucleic acid (rDNA) 16s and the second directed to confirm C. acnes through specific rDNA 16s primers.
  Arms: Phenotypic and genotypic characterization
Genetic: Multiomics analysis — Whole Genome Sequencing, proteomics and metabolomics analysis
  Arms: Multiomics analysis

SUMMARY:
The study aims to identify metabolites present in intervertebral discs colonized by C. acnes from patients with low back pain and degenerative disc disease, correlating them with their clinical, radiological and demographic profiles.

ELIGIBILITY:
Inclusion Criteria:

* low back pain lasting longer than 3 months;
* MRI findings of degenerative lumbar discopathy (DDL) performed less than 6 months after inclusion in the study;
* indication for open surgical treatment, with isolated microdiscectomy or associated with lumbar arthrodesis;
* failure of conservative treatment for at least 6 weeks and/or progressive neurological deficit

Exclusion Criteria:

* History of open lumbar spine surgery at any stage of life;
* presence of chemotherapy or pulse therapy with corticoids;
* patients with immune deficiency;
* patients undergoing previous intradiscal therapies (nucleotomy or discography);
* patients undergoing previous endoscopic surgery;
* patients with a history of previous spinal infection treated with antibiotics in the 6 months prior to inclusion in the study;
* use of antibiotics in the 2 months prior to the surgical procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of C. acnes on intervertebral disc | Up to 5 months
  Incidence of C. acnes on intervertebral disc in patients with chronic low back pain and DDL.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitário Gaffrée e Guinle, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Magno da Rocha V, Lima COGX, Ferreira EO, de Farias GC, Nogueira FCS, Martha Antunes LC, Cassiano KM, Fiorelli RKA. Colonization of intervertebral discs by Cutibacterium acnes in patients with low back pain: Protocol for an analytical study with microbiological, phenotypic, genotypic, and multiomic techniques. PLoS One. 2023 Feb 27;18(2):e0271773. doi: 10.1371/journal.pone.0271773. eCollection 2023. PMID 36848344